CLINICAL TRIAL: NCT00078377
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of CEP-10953 (150 and 250 mg/Day) as Treatment for Adults With Excessive Sleepiness Associated With Narcolepsy
Brief Title: Safety and Efficacy Study of Armodafinil (CEP-10953) in the Treatment of Excessive Sleepiness Associated With Narcolepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/3020/NA/MN
Record Dates: First submitted 2004-02-24; First posted 2004-02-26 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Excessive Sleepiness; Cataplexy; Sleep Attacks; Excessive Sleepiness associated with Narcolepsy; Cephalon; Cephalon, Inc; Nuvigil
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Cataplexy | interventions — Modafinil

ARMS (3):
- 1 (Experimental): Armodafinil 250 mg
  Interventions: Drug: Armodafinil
- 2 (Experimental): Armodafinil 150 mg
  Interventions: Drug: Armodafinil
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Armodafinil 250 mg once daily in the morning
  Arms: 1
Drug: Armodafinil — Armodafinil 150 mg once daily in the morning
  Arms: 2
Drug: Placebo — Matching placebo tablets once daily
  Arms: 3

SUMMARY:
The primary objective of this study is to determine whether treatment with Armodafinil (CEP-10953) is more effective than placebo treatment for patients with excessive sleepiness associated with narcolepsy by measuring mean sleep latency from the Maintenance of Wakefulness Test (MWT) (20-minute version)(average of 4 naps at 0900, 1100, 1300, and 1500) and by the Clinical Global Impressions of Change (CGI-C) ratings (as related to general condition) at week 12 (or last postbaseline observation)

ELIGIBILITY:
Diagnosis and Criteria for Inclusion:

Patients are included in the study if all of the following criteria are met:

* Written informed consent is obtained
* The patient is an outpatient, man or woman of any ethnic origin, 18 to 65 years of age (inclusive)
* The patient has a complaint of excessive sleepiness
* The patient has a current diagnosis of narcolepsy according to ICSD criteria.
* The patient is in good health as determined by a medical and psychiatric history, physical examination, electrocardiogram (ECG), and serum chemistry, hematology, and urinalysis.
* Women must be surgically sterile, 2 years postmenopausal, or, if of child-bearing potential, using a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]) and agree to continued use of this method for the duration of the study.
* The patient has a mean sleep latency of 6 minutes or less as determined by the Multiple Sleep Latency Test (MSLT) (performed at 0900, 1100, 1300, and 1500).
* The patient has a CGI-S (Clinical Global Impression of Severity of Illness) rating of 4 or more.
* The patient does not have any medical or psychiatric disorders that could account for the excessive daytime sleepiness.
* The patient is able to complete self rating scales and computer-based testing.
* The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Criteria for Exclusion:

Patients are excluded from participating in this study if 1 or more of the following criteria are met. The patient:

* has any clinically significant, uncontrolled medical or psychiatric conditions (treated or untreated)
* has a probable diagnosis of a current sleep disorder other than narcolepsy
* consumed caffeine including coffee, tea and/or other caffeine containing beverages or food averaging more than 600 mg of caffeine per day
* used any prescription drugs disallowed by the protocol or clinically significant use of over the-counter (OTC) drugs within 7 days before the second screening visit
* has a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM IV)
* has a positive UDS at the screening visit, without medical explanation
* has a clinically significant deviation from normal in the physical examination
* is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
* has used an investigational drug within 1 month before the screening visit
* has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery)
* has a known clinically significant drug sensitivity to stimulants or modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 centers in the US, Canada, France, Germany, Russia, and Australia. First patient enrolled (treatment): 23 March 2004/ Last patient last visit: 10 January 2005
Pre-assignment Details: 2 female patients withdrew after randomization but prior to receiving study drug (1 withdrew consent and 1 was lost to follow-up)
Groups:
- Armodafinil 250 mg/Day: Armodafinil 250 mg once daily in the morning
- Armodafinil 150 mg/Day: Armodafinil 150 mg once daily in the morning
- Placebo: Matching placebo tablets once daily in the morning
Period: Overall Study
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Started | 67 | 65 | 64
Completed | 56 | 49 | 55
Not Completed | 11 | 16 | 9
Not completed — Adverse Event | 2 | 5 | 1
Not completed — Lack of Efficacy | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 4
Not completed — Miscellaneous | 2 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 67 | 65 | 64 | 196
Age Categorical [Number; unit: participants] — 2 female patients withdrew after randomization but prior to receiving study drug (1 withdrew consent and 1 was lost to follow-up)
  participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 66 | 64 | 63 | 193
    >=65 years | 1 | 0 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 35.0 (12.52) | 40.4 (12.52) | 39.2 (11.98) | 38.1 (12.50)
Gender [Number; unit: participants] — 2 female patients withdrew after randomization but prior to receiving study drug (1 withdrew consent and 1 was lost to follow-up)
  participants
    Female | 42 | 36 | 31 | 109
    Male | 25 | 28 | 32 | 85
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 37 | 111
  Canada | 12 | 12 | 12 | 36
  France | 3 | 3 | 3 | 9
  Germany | 5 | 4 | 4 | 13
  Russian Federation | 5 | 4 | 4 | 13
  Australia | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maintenance of Wakefullness Test (MWT) Score at 12 Weeks
Description: The Maintenance of Wakefulness Test (MWT) is an objective assessment of sleepiness that measures the ability of a subject to remain awake. Long latencies to sleep are indicative of a patient's ability to remain awake. The change from baseline in the mean sleep latency from the MWT (average of 4 tests at 0900, 1100, 1300, and 1500) was analyzed at weeks 4, 8, and 12. The primary efficacy variable was the mean change from the baseline assessment in MWT sleep latency as assessed at week 12 (or last post-baseline visit).
Time Frame: change from baseline at 12 weeks
Population: Safety Analysis set of 194 total patients: 2 patients withdrew after randomization but prior to receiving study drug (1 withdrew consent and 1 was lost to follow-up).
  Full Analysis set of 176 total patients: 18 patients that had withdrawn from the study were non-evaluable for efficacy.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo | Armodafinil Combined Group (250 mg/Day and 150 mg/Day)
Number analyzed (Participants) | 60 | 58 | 58 | 118
Minutes | 2.6 (6.24) | 1.3 (6.31) | -1.9 (6.87) | 1.9 (6.28)
Statistical Analysis 1: Comparison: Armodafinil 250 mg/Day vs Armodafinil 150 mg/Day vs Placebo; Statistical data is for the Armodafinil Combined treatment (250 mg/day and 150 mg/day groups) compared to the placebo treatment group; Test type: Superiority or Other; p = 0.0024, ANCOVA; The corresponding baseline value as a covariate; Mean Difference (Final Values) = 3.8, 95% CI [1.02 to 4.61]

2. Primary Outcome: Change From Baseline in Clinical Global Impression of Change (CGI-C) Score at 12 Weeks
Description: Number of participants who had at least minimal improvement in CGI-C ratings at Week 12 or last post-baseline visit. The CGI-C uses the following categories and scoring assignments: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; and 7=Very much worse. Severity of illness was assessed at baseline by the CGI-S, which consists of the following categories: 1=Normal (shows no signs of illness); 2=Borderline ill; 3=Mildly (Slightly) ill; 4=Moderately ill; 5=Markedly ill; 6=Severely ill; and 7=Among the most extremely ill patients.
Time Frame: change from baseline at 12 weeks
Population: Safety Analysis set of 194 total patients (received at least 1 dose of study drug): 2 patients withdrew after randomization but prior to receiving study drug (1 withdrew consent and 1 was lost to follow-up).
  Full Analysis set of 176 total patients: 18 patients that had withdrawn from the study were non-evaluable for efficacy analysis.
Measure: Number; unit: Participants
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo | Armodafinil Combined Group (250 mg/Day and 150 mg/Day)
Number analyzed (Participants) | 60 | 58 | 58 | 118
Participants | 60 | 58 | 58 | 118
Statistical Analysis 1: Comparison: Placebo vs Armodafinil Combined Group (250 mg/Day and 150 mg/Day); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Armodafinil 250 mg/Day | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/64 | 0/63
Other Adverse Events (participants affected / at risk) | 29/67 | 21/64 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 250 mg/Day (N=67) | Armodafinil 150 mg/Day (N=64) | Placebo (N=63)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 250 mg/Day (N=67) | Armodafinil 150 mg/Day (N=64) | Placebo (N=63)
Nausea (Gastrointestinal disorders) | 5 | 9 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 0
Headache (Nervous system disorders) | 19 | 10 | 7
Dizziness (Nervous system disorders) | 2 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days